CLINICAL TRIAL: NCT03210272
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 1358894 in Healthy Male Subjects (Single-blind, Partially Randomised, Placebo-controlled Parallel Group Design) and Effect of Food on the Relative Bioavailability of BI 1358894 (Open-label, Randomised, Two-way Cross-over)
Brief Title: This Study in Healthy Men Tests How Different Doses of BI 1358894 Are Taken up in the Body and How Well They Are Tolerated. The Study Also Looks at How Food Influences the Amount of BI 1358894 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1402-0001; 2017-000143-40 (EudraCT Number)
Record Dates: First submitted 2017-07-05; First posted 2017-07-06 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — TRPC inhibitor BI 1358894

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single rising dose part (Experimental): Group of healthy male volunteers receive rising single doses of BI 1358894
  Interventions: Drug: Placebo; Drug: BI 1358894
- Food effect part (Experimental): Group of healthy male volunteers receive single doses of BI 1358894 with and without food
  Interventions: Drug: BI 1358894 (Test); Drug: BI 1358894 (Reference)

INTERVENTIONS:
Drug: Placebo — Tablet
  Arms: Single rising dose part
Drug: BI 1358894 — Tablet
  Arms: Single rising dose part
Drug: BI 1358894 (Test) — Fasting state
  Arms: Food effect part
Drug: BI 1358894 (Reference) — Fed state
  Arms: Food effect part

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 1358894 in healthy male subjects following oral administration of single rising doses. Secondary objectives are the exploration of the pharmacokinetics (PK), including dose proportionality of BI 1358894 after single dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 45 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
* Willingness to comply with contraception requirements. Subjects who are sexually active, must use, with their female partner, adequate contraception throughout the study and until one month after the last administration of trial medication. Adequate methods are:

  * Sexual abstinence or
  * A vasectomy performed at least 1 year prior to screening in combination with a barrier method (condom) or
  * Surgical sterilisation (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy) of the subjects female partner or
  * The use of condoms, if the female partner uses in addition an adequate contraception method, e.g., intrauterine device (IUD), hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to first drug administration, or barrier method (e.g. diaphragm with spermicide)
* Unprotected sexual intercourse with a pregnant female partner is not allowed throughout the study and until one month after the last administration of trial medication

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* C-Reactive Protein > ULN, erythrocyte sedimentation rate (ESR) ≥ 15 millimeters/hour, liver and kidney parameter above ULN, other laboratory values outside the reference range the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more 30 g per day for males)
* Drug abuse as per investigator judgment or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Any lifetime history of suicidal behaviour (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behaviour)
* Any suicidal ideation of type 2 to 5 on the C-SSRS in the past 12 months (i.e. active suicidal thought, active suicidal thought with method, active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fuertig R, Goettel M, Herich L, Hoefler J, Wiebe ST, Sharma V. Effects of Single and Multiple Ascending Doses of BI 1358894 in Healthy Male Volunteers on Safety, Tolerability and Pharmacokinetics: Two Phase I Partially Randomised Studies. CNS Drugs. 2023 Dec;37(12):1081-1097. doi: 10.1007/s40263-023-01041-4. Epub 2023 Nov 29. PMID 38019355

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single rising oral doses of BI 1358894 in healthy male subjects (single-blind, partially randomised, placebo-controlled parallel group design) and effect of food on the relative bioavailability of BI 1358894 (open-label, randomised, two-way cross-over)
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they met all implemented inclusion/exclusion criteria, Subjects were not to be randomised to trial drug if any of the specific entry criteria was violated
Groups:
- Placebo: matching placebo Single Rising Dose (SRD) part
- BI 3mg: oral administration of BI 1358894 film-coated tablet (3*1 milligram (mg) tablet) Single Rising Dose (SRD) part
- BI 6mg: oral administration of BI 1358894 film-coated tablet (6*1mg tablet) Single Rising Dose (SRD) part
- BI 10mg: oral administration of BI 1358894 film-coated tablet (2*5mg tablet) Single Rising Dose (SRD) part
- BI 25mg: oral administration of BI 1358894 film-coated tablet (1*25mg tablet) Single Rising Dose (SRD) part
- BI 50mg: oral administration of BI 1358894 film-coated tablet (2*25mg tablet) Single Rising Dose (SRD) part
- BI 100mg: oral administration of BI 1358894 film-coated tablet (1*100mg tablet) Single Rising Dose (SRD) part
- BI 200mg Fast: oral administration of BI 1358894 film-coated tablet in fasting status (2*100mg tablet) Single Rising Dose (SRD) part
- BI 200mg Fed: oral administration of BI 1358894 film-coated tablet in fed status (2*100mg tablet) Single Rising Dose (SRD) part
- BI 50mg Fed / BI 50mg Fast: oral administration of BI 1358894 film-coated tablet in fed state (Test) (2*25mg)/ oral administration of BI 1358894 film-coated tablet in fasting state (Reference) (2*25mg) Food effect (FE) part
- BI 50mg Fast / BI 50m Fed: oral administration of BI 1358894 film-coated tablet in fasting state (Reference) (2*25mg) / oral administration of BI 1358894 film-coated tablet in fed state (Test) (2*25mg) Food effect (FE) part
- BI 100mg Fed / BI 100mg Fast: oral administration of BI 1358894 film-coated tablet in fed state (Test) (1*100mg)/ oral administration of BI 1358894 film-coated tablet in fasting state (Reference) (1*100mg) Food effect (FE) part
- BI 100mg Fast / BI 100m Fed: oral administration of BI 1358894 film-coated tablet in fasting state (Reference) (1*100mg)/ oral administration of BI 1358894 film-coated tablet in fed state (Test) (1*100mg) Food effect (FE) part
Period: Overall Study
Arm/Group | Placebo | BI 3mg | BI 6mg | BI 10mg | BI 25mg | BI 50mg | BI 100mg | BI 200mg Fast | BI 200mg Fed | BI 50mg Fed / BI 50mg Fast | BI 50mg Fast / BI 50m Fed | BI 100mg Fed / BI 100mg Fast | BI 100mg Fast / BI 100m Fed
Started | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 4 | 6 | 6
Completed | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 4 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS):
  This subject set included all subjects who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 3mg | BI 6mg | BI 10mg | BI 25mg | BI 50mg | BI 100mg | BI 200mg Fast | BI 200mg Fed | BI 50mg Fed / BI 50mg Fast | BI 50mg Fast / BI 50m Fed | BI 100mg Fed / BI 100mg Fast | BI 100mg Fast / BI 100m Fed | Total
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 4 | 6 | 6 | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.7 (5.8) | 40.2 (7.4) | 33.7 (7.4) | 36.2 (6.0) | 36.2 (7.3) | 40.2 (3.5) | 35.5 (6.6) | 38.3 (7.0) | 28.0 (3.6) | 36.8 (8.8) | 32.5 (8.3) | 34.2 (10.2) | 30.0 (8.1) | 34.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 4 | 6 | 6 | 83
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  White | 15 | 6 | 5 | 6 | 5 | 6 | 6 | 6 | 5 | 4 | 4 | 6 | 6 | 80
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug- Related Adverse Event
Description: Percentage of subjects with drug-related adverse events
Time Frame: From start of treatment until end of trial. Up to 14 days for single rising dose part under fasting condition (3mg to 200mg) and the food effect part and up to 33 days for the single rising dose part under fed conditions (200mg fed dose group)
Population: as for baseline characteristics
Measure: Number; unit: Percentage
Groups:
- BI 50mg Fed: oral administration of BI 1358894 film-coated tablet in fed state (Test) (2*25mg), Food effect (FE) part
- BI 50mg Fast: oral administration of BI 1358894 film-coated tablet in fasting state (Reference) (2*25mg), Food effect (FE) part
- BI 100mg Fed: oral administration of BI 1358894 film-coated tablet in fed state (Test) (1*100mg), Food effect (FE) part
- BI 100mg Fast: oral administration of BI 1358894 film-coated tablet in fasting state (Reference) (1*100mg), Food effect (FE) part
Arm/Group | Placebo | BI 3mg | BI 6mg | BI 10mg | BI 25mg | BI 50mg | BI 100mg | BI 200mg Fast | BI 200mg Fed | BI 50mg Fed | BI 50mg Fast | BI 100mg Fed | BI 100mg Fast
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 12 | 12
Percentage | 0.0 | 16.7 | 50.0 | 0.0 | 33.3 | 66.7 | 66.7 | 50.0 | 66.7 | 87.5 | 87.5 | 50.0 | 66.7

2. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte BI1358894 in Plasma Over the Time Interval From 0 Extrapolated to Infinity
Description: Area under the concentration-time curve of the analyte BI1358894 in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf)
Time Frame: Within 2 hours (h) before and 0.167h, 0.333h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 16h, 24h, 36h, 48h, 72h, 96h, 120h, 144h, 192h after drug administration
Population: Pharmacokinetic parameter analysis set (PKS):
  The PK parameter analysis set (PKS) included all subjects from the TS receiving BI 1358894 who provided at least 1 secondary PK parameter (AUC or Cmax) that was not excluded because of protocol deviations relevant to the statistical evaluation of PK endpoints
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles*Hour per Litre
Groups:
- BI 50mg Fast (R): oral administration of BI 1358894 film-coated tablet (2*25mg tablet) in fasting status (Reference) Food effect (FE) part
- BI 50 mg Fed (T): oral administration of BI 1358894 film-coated tablet (2*25mg tablet) in fed status (Test) Food effect part
- BI 100mg Fast (R): oral administration of BI 1358894 film-coated tablet (1*100 mg tablet) in fasting status (Reference) Food effect part
- BI 100mg Fed (T): oral administration of BI 1358894 film-coated tablet (1*100 mg tablet) in fed status (Test) Food effect (FE) part
Arm/Group | BI 3mg | BI 6mg | BI 10mg | BI 25mg | BI 50mg | BI 100mg | BI 200mg Fast | BI 200mg Fed | BI 50mg Fast (R) | BI 50 mg Fed (T) | BI 100mg Fast (R) | BI 100mg Fed (T)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 12 | 12
Nanomoles*Hour per Litre | 341 (20.7) | 596 (33.3) | 922 (20.4) | 2540 (29.9) | 4470 (25.5) | 2960 (1570) | 13700 (45.7) | 33800 (30.1) | 4920 (27.1) | 7660 (41.0) | 7020 (56.4) | 16900 (21.5)
Statistical Analysis 1: Comparison: BI 50mg Fast (R) vs BI 50 mg Fed (T); The statistical model to assess relative bioavailability in the FE part was an analysis of variance (ANOVA) on the ln-transformed parameters AUC and Cmax including effects for 'sequence', 'subjects nested within sequences', 'period', and 'treatment'; Test type: Other; Geometric Mean Ratio T/R (%) = 155.60, 90% CI 2-sided [130.66 to 185.30] — intra-individual gCV (%) = 18.1
Statistical Analysis 2: Comparison: BI 100mg Fast (R) vs BI 100mg Fed (T); [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratio T/R (%) = 240.12, 90% CI 2-sided [196.25 to 293.81] — intra-individual gCV (%) = 27.8

3. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte BI1358894 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Time Point
Description: Area under the concentration-time curve of the analyte BI1358894 in plasma over the time interval from 0 to the last quantifiable data time point (AUC0-tz).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles*Hour per Litre
Arm/Group | BI 3mg | BI 6mg | BI 10mg | BI 25mg | BI 50mg | BI 100mg | BI 200mg Fast | BI 200mg Fed | BI 50mg Fast (R) | BI 50 mg Fed (T) | BI 100mg Fast (R) | BI 100mg Fed (T)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 12 | 12
Nanomoles*Hour per Litre | 288 (18.5) | 569 (32.7) | 861 (17.7) | 2380 (29.7) | 4170 (26.2) | 2520 (2670) | 12600 (42.0) | 32800 (29.0) | 4440 (23.5) | 6940 (36.2) | 6320 (53.4) | 15500 (19.3)
Statistical Analysis 1: Comparison: BI 50mg Fast (R) vs BI 50 mg Fed (T); [analysis description as in outcome 2, analysis 1]; Test type: Other; Geometric Mean Ratio T/R (%) = 156.37, 90% CI 2-sided [132.73 to 184.22] — intra-individual gCV (%) = 17.0
Statistical Analysis 2: Comparison: BI 100mg Fast (R) vs BI 100mg Fed (T); [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratio T/R (%) = 245.56, 90% CI 2-sided [200.70 to 300.44] — intra-individual gCV (%) = 27.8

4. Secondary Outcome: Maximum Measured Concentration of the Analyte BI 1358894 in Plasma
Description: Maximum measured concentration of the analyte BI 1358894 in plasma (Cmax).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles per Litre
Arm/Group | BI 3mg | BI 6mg | BI 10mg | BI 25mg | BI 50mg | BI 100mg | BI 200mg Fast | BI 200mg Fed | BI 50mg Fast (R) | BI 50 mg Fed (T) | BI 100mg Fast (R) | BI 100mg Fed (T)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 12 | 12
Nanomoles per Litre | 27.6 (30.0) | 35.9 (33.8) | 59.7 (13.4) | 84.2 (44.2) | 183 (56.3) | 94.3 (735) | 385 (26.8) | 857 (22.2) | 149 (59.4) | 237 (24.9) | 210 (38.8) | 517 (8.61)
Statistical Analysis 1: Comparison: BI 50mg Fast (R) vs BI 50 mg Fed (T); [analysis description as in outcome 2, analysis 1]; Test type: Other; Geometric Mean Ratio T/R (%) = 158.74, 90% CI 2-sided [114.25 to 220.56] — intra-individual gCV (%) = 34.8
Statistical Analysis 2: Comparison: BI 100mg Fast (R) vs BI 100mg Fed (T); [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratio T/R (%) = 246.13, 90% CI 2-sided [203.37 to 297.89] — intra-individual gCV (%) = 26.2

ADVERSE EVENTS:
Time Frame: From start of treatment until end of trial. Up to 14 days for single rising dose part under fasting condition (3mg to 200mg) and the food effect part and up to 33 days for the single rising dose part under fed conditions (200mg fed dose group)
Description: Treated set (TS): This subject set included all subjects who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment.
Groups:
- BI Total SRD: total summary BI 1358894
- BI 50mg Fed: oral administration of BI 1358894 film-coated tablet (2*25mg tablet) in fed status (Test) Food effect (FE) part
- BI 100mg Fast (R): oral administration of BI 1358894 film-coated tablet (1*100 mg tablet) in fasting status (Reference) Food effect (FE) part
Arm/Group | Placebo | BI 3mg | BI 6mg | BI 10mg | BI 25mg | BI 50mg | BI 100mg | BI 200mg Fast | BI 200mg Fed | BI Total SRD | BI 50mg Fed | BI 50mg Fast (R) | BI 100mg Fed (T) | BI 100mg Fast (R)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/48 | 0/8 | 0/8 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/48 | 0/8 | 0/8 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/15 | 3/6 | 6/6 | 0/6 | 2/6 | 4/6 | 4/6 | 3/6 | 6/6 | 28/48 | 7/8 | 7/8 | 6/12 | 8/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | BI 3mg (N=6) | BI 6mg (N=6) | BI 10mg (N=6) | BI 25mg (N=6) | BI 50mg (N=6) | BI 100mg (N=6) | BI 200mg Fast (N=6) | BI 200mg Fed (N=6) | BI Total SRD (N=48) | BI 50mg Fed (N=8) | BI 50mg Fast (R) (N=8) | BI 100mg Fed (T) (N=12) | BI 100mg Fast (R) (N=12)
Auditory disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 3 | 2 | 3
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 4 | 0 | 2 | 3 | 3 | 3 | 3 | 20 | 6 | 7 | 4 | 7
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Apathy (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT03210272/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT03210272/SAP_001.pdf